CLINICAL TRIAL: NCT07227389
Title: The Relationship Between Timing of Opioid Administration and Postoperative Respiratory Depression.
Brief Title: Timing of Opioid Administration and Postoperative Respiratory Depression.
Status: Not yet recruiting | Type: Observational
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Wael Saasouh, MD, Clinical Assistant Professor, Wayne State University
Other Study IDs: IRB-23-08-6045
Record Dates: First submitted 2025-11-07; First posted 2025-11-12 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Respiratory Complications; Opioid Induced Respiratory Depression; Postoperative Respiratory Complications
Keywords: opioids; bio-impedance; hypoxia; hypercapnia; minute ventilation
MeSH Terms: conditions — Hypoxia; Hypercapnia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients receiving general anesthesia with an expected anesthetic time of at least 2 hours
  Interventions: Diagnostic Test: Respiratory volume monitoring

INTERVENTIONS:
Diagnostic Test: Respiratory volume monitoring — Noninvasive continuous respiratory monitoring utilizing bio-impedance to detect tidal volumes, respiratory rate, and minute ventilation.

SUMMARY:
The goal of this study is to determine if a relationship can be detected between the administration of an opioid and quantitative respiratory depression in spontaneously breathing non-intubated patients who have undergone general anesthesia and have received perioperative opioids.

The primary aim is to determine the temporal effect of opioid administration on respiratory depression as assessed by minute ventilation with a reduction of at least 20% in the percent of predicted minute ventilation.

A secondary aim is to determine a dose response of opioid administration and its effect on minute ventilation.

The investigators aim to determine the influence of opioid administration on minute ventilation on spontaneously breathing patients during post-anesthesia care unit (PACU) stay.

DETAILED DESCRIPTION:
Opioids have been used as a mainstay of perioperative analgesia since the late 18th century. The use of opioids, however, is not without risk as both short-term and long-term complications have been reported leading to in-hospital morbidity as well as increased 30-day readmission. Multiple postoperative complications are attributed to opioid administration including respiratory, cardiovascular, neurological, and gastrointestinal. As such, the routine use of opioids postoperatively is constantly being re-evaluated in search of better alternatives. For the time being, opioid prescription is largely provider dependent and hence the complications are varied. Opioids act on central and peripheral receptors leading to analgesia, but also cause worsening sleep apnea, decreased ventilatory response to hypoxia and hypercarbia, and may lead to hyperalgesia and sedation, thus feeding a vicious cycle. Certain patient populations have increased analgesic demand postoperatively and are thus at increased risk of postoperative opioid-induced respiratory depression (OIRD). This is especially true in patients with morbid obesity, chronic opioid use, obstructive sleep apnea (OSA), or sleep-disordered breathing (SDB). Higher risk patients also include those with concomitant pulmonary disease. The morbidity and mortality are even higher in the unmonitored setting. Current efforts at monitoring postoperative patients are mostly intermittent peripheral oximetry checks by the inpatient ward staff unless the patient is present in a step-down or intensive care unit. There are no clear guidelines on continuous postoperative oxygenation monitoring mostly due to the lack of published data. Intermittent checks are typically done every four or eight hours and are generally suboptimal at detecting episodes of hypoxemia. Other indirect methods of measuring hypoxemia include incidence of naloxone administration and/or code blue (cardio-respiratory arrest) emergencies. While continuous peripheral pulse oximetry in the postoperative period is currently the best available means to detect hypoxemia, it is not without flaws. Several factors can lead to falsely decreased measured oxygen saturation including motion artifacts, cold fingers, and sleep position. Oximetry would also detect hypoxemia after the oxygen reserves have been depleted, which is usually later in the process. Most preventable deaths attributable to OIRD seem to occur shortly after release from the post-anesthesia care unit (PACU) and are more likely during the night shift or during other times of decreased nursing availability. Noninvasive continuous respiratory monitoring is possible using a novel respiratory volume monitor (RVM) that utilizes bio-impedance to detect tidal volumes, respiratory rate, and minute ventilation in non-intubated patients (ExSpiron). The realtime minute ventilation (MV) as obtained from the RVM is contrasted with the calculated predicted MV according to the patients size and gender to end up with a percent of the predicted MV (%MVPRED) that relates to the degree of respiratory depression. The use and quantification of this ratio can aid in analyzing the respiratory effect that an opioid dose can have on the patient. Where a MVPRED of 80% can relate to mild respiratory depression. Here the investigators aim to capture the influence of opioid dosage on minute ventilation, with a primary outcome of a %MVPRED reduction of at least 20%. Respiratory Metrics: Respiratory metrics, including MV, %MVPRED, TV, and RR will be recorded by the Respiratory Volume Monitor (ExSpiron, Senzime, Uppsala, Sweden). Metrics will be recorded every 5 seconds and calculated as an average of the previous 30-second window. De-identified respiratory metric data will be downloaded directly from each patient every day and at the completion of the study using the built-in user interface. Clinicians will be asked to record the precise time of any respiratory interventions.

Rationale for conducting the research: The researchers propose to evaluate the effect of opioids on respiratory depression as monitored by a non-invasive respiratory volume monitor on postoperative non-intubated patients. Primarily, the aim is to determine the correlation between opioid administration and decreased respiratory function. More specifically, the immediate effect that opioid administration has on minute ventilation. In order to test this relationship, the researchers put forward a blinded observation study on adult patients in the PACU who require pain management with opioids.

Rationale for the selected participant population: Patients in the PACU often require pain management with opioids. Monitoring these patients with a non-invasive respiratory monitor for opioid induced respiratory depression (OIRD) may potentially detect adverse events earlier than conventional standard of care monitors.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Adults ≥18 years of age and ≤85 years of age
* Patients planned for general anesthesia with an expected anesthetic time of at least 2 hours
* Patients expected to receive postoperative opioid analgesia

Exclusion Criteria:

* Non-operative procedure (imaging)
* Patients not admitted to the PACU postoperatively
* Use of patient-controlled analgesia systems
* Female patients who are pregnant or breastfeeding
* Patients with asymmetric lung disease
* American Society of Anesthesiologists (ASA) classification V
* Emergency surgery (ASA E Modifier)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Surgical patients receiving general anesthesia with an expected anesthetic time of at least 2 hours
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Respiratory interventions 1 | Within 4 hours of patient admittance to Post Anesthetic Care Unit (PACU)
  Initiation or cessation of mechanical ventilation
Respiratory interventions 2 | Within 4 hours of patient admittance to Post Anesthetic Care Unit
  Initiation or cessation of Bilevel Positive Airway Pressure
Respiratory interventions 3 | Within 4 hours of patient admittance to Post Anesthetic Care Unit
  Initiation/cessation of high flow nasal cannula
Respiratory interventions 4 | Within 4 hours of patient admittance to Post Anesthetic Care Unit
  Initiation/cessation of low flow nasal cannula

SECONDARY OUTCOMES:
Oxygen saturation of peripheral blood (SpO2) | Duration of PACU stay (up to 4 hours)
  Oxygen saturation of peripheral blood during PACU stay
Arterial Blood gas levels | Duration of surgery (up to 2hrs)
  Arterial Blood gas levels during surgery
Venous Blood gas levels | Duration of surgery (up to 2hrs)
  Venousl Blood gas levels during surgery
Hypercapnia | Duration of patient stay in PACU (up to 4 hours)
  Hypercapnic episode as measured by EtCO2
Hypoxia | Duration of patient stay in PACU (up to 4 hours)
  Hypoxic episodes episode as measured by SpO2
Patient transfer occurrence | During patient stay (up to 30 days)
  Patient transfer to higher/lower acuity level such as ICU, hospital floor, step-down unit
Initiation of patient prone position placement | During patient PACU stay (up to 4 hours)
  Occurance time of patient placement into the prone position

CONTACTS AND LOCATIONS:
Overall Officials: Wael Saasouh, MD, Principal Investigator — Wayne State University
Locations (1):
- Detroit Medical Center, Mount Clemens, Michigan, United States

IPD SHARING:
Plan to Share IPD: No